CLINICAL TRIAL: NCT05760066
Title: Effects of Resistance Training Preconditioning on Skeletal Muscle Recovery From a Period of Disuse in Young Adults
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Auburn University (Other)
Responsible Party: Principal Investigator, Michael Roberts, Professor, Auburn University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MDR0823
Record Dates: First submitted 2023-01-23; First posted 2023-03-08 (Actual); Last update posted 2023-03-08 (Actual); Status verified 2023-02

CONDITIONS: Atrophy, Disuse; Atrophy, Muscular
MeSH Terms: conditions — Muscular Disorders, Atrophic; Muscular Atrophy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Resistance Training Preconditioning (PRECON) (Experimental): This group will perform:
  1. 6 weeks of lower body focused resistance training
  2. 2 weeks of locking brace-induced immobilization of a randomized leg
  3. 6 weeks of lower body focused resistance training
  Interventions: Other: Resistance Training Preconditioning
- Control (CTL) (Active Comparator): This group will perform:
  1. 6 weeks of activities of daily living (no training)
  2. 2 weeks of locking brace-induced immobilization of a randomized leg
  3. 6 weeks of lower body focused resistance training
  Interventions: Other: Control

INTERVENTIONS:
Other: Resistance Training Preconditioning — Resistance training prior to disuse-induced atrophy followed by another period of resistance training
  Arms: Resistance Training Preconditioning (PRECON)
Other: Control — Activities of daily living prior to disuse-induced atrophy followed by a period of resistance training
  Arms: Control (CTL)

SUMMARY:
The goal of this clinical trial is to compare the effects of resistance training (RT) preconditioning vs no training on disuse-induced atrophy and post-disuse resistance training in young healthy individuals. The main questions it aims to answer are:

* To determine if performing RT prior to a period of disuse enhances the regain of strength, skeletal muscle size, and skeletal muscle quality while performing RT after a period of disuse.
* To determine if performing RT prior to a period of disuse dampens the maladaptive effects of disuse on muscle size, muscle quality, and strength.
* To determine the anabolic and proteolytic mechanisms underpinning the observed outcomes.

Participants will:

1. Perform either 6 weeks of resistance training or maintain an untrained lifestyle
2. Perform 2 weeks of limb immobilization induced disuse of a randomized leg
3. Perform 6 weeks of resistance training

Researchers will compare the resistance training preconditioning condition vs the non-trained condition to see if resistance training prior to a period of disuse is beneficial during the disuse period and in the return to training period on skeletal muscle size, strength, and underpinning molecular markers.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18-30
* Free from medical implants in lower extremity that would interfere with low-dose radiation
* Are not allergic to ultrasound gel or Lidocaine
* Have no or minimal experience with resistance training (less than 1 training session/week for a 1 year period)

Exclusion Criteria:

* Have been exposed to medically necessary radiation in the past 12 months other than dental x-rays
* Have known overt cardiovascular or metabolic disease
* Have a medical condition that would contraindicate participating in an exercise program or donating a skeletal muscle biopsy (e.g. blood clotting disorder, taking blood thinners, etc.)
* Are undergoing medical treatment for a disease that would interfere physiologically or logistically with study outcomes and/or protocols (e.g. undergoing chemotherapy and/or radiation for cancer treatment)
* Have consumed supplemental protein, creatine, and/or agents that affect hormone status (e.g. testosterone, growth hormone boosters, etc.) within the previous 2 months.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2023-08-01 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-08-01 (Estimated)

PRIMARY OUTCOMES:
Change in vastus lateralis fiber cross-sectional area | Through completion of study, 16 weeks
  Upon the procurement and analysis of muscle from the vastus lateralis of participants, histological techniques will be used to assess fiber cross-sectional area of muscle fibers
Change in quadriceps strength via 3 repetition maximum testing | Through completion of study, 16 weeks
  Strength of the quadriceps will be assessed via 3-repetition maximum testing of select exercises (leg press, leg extension, hex-bar deadlift)
Change in quadriceps strength via isokinetic dynamometry | Through completion of study, 16 weeks
  Strength of the quadriceps will be assessed via isokinetic dynamometry

SECONDARY OUTCOMES:
Change in protein expression of anabolic signaling proteins | Through completion of study, 16 weeks
  Western blotting will be performed and quantified in relative fluorescence units for proteins involved in the mechanistic target of rapamycin signaling pathway.
Change in protein expression of catabolic signaling proteins | Through completion of study, 16 weeks
  Western blotting will be performed and quantified in relative fluorescence units for proteins involved in the catabolic signaling pathways (e.g. ubiquitin-proteasome system, calpain system, autophagy).
Change in activity of catabolic systems | Through completion of study, 16 weeks
  Activity assays will be performed and quantified in relative fluorescence units normalized to muscle soluble protein abundance in order to quantify the activity of the calpain system and the 20S proteasome core.
Gene expression at the mRNA level of atrophy-associated genes (atrogenes) | Through completion of study, 16 weeks
  Real time quantitative polymerase chain reactions (qPCR) will be used to quantify the expression of select genes associated with atrophy. These data will be reported as fold-change from baseline and will be normalized to one or more housekeeping genes whose value does not change throughout the duration of the study.